CLINICAL TRIAL: NCT02873429
Title: Measuring the Context of Healing: Using PROMIS in Chronic Pain Treatment
Brief Title: Measuring the Context of Healing in Chronic Pain Treatment
Acronym: HEALpain
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Carol Greco, Associate Professor of Psychiatry, University of Pittsburgh
Other Study IDs: ME-1402-10114
Record Dates: First submitted 2016-08-12; First posted 2016-08-19 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-04

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Integrative Medicine (Complementary /Alternative)Group: Patients receiving chiropractic care, acupuncture, massage therapy, or meditation training for chronic pain
- Conventional Medicine Group: Patients receiving conventional medicine care (physical therapy, medication management, injections, etc.) for chronic pain.

SUMMARY:
This project focuses on whether nonspecific factors as well as patient characteristics contribute to treatment outcome differences. The project uses assessment instruments, computerized adaptive tests (CATs), from the Patient-Reported Outcomes Measurement Information System (PROMIS®). The research team has recently developed and tested (using PROMIS methods) a set of instruments to assess non-specific factors in healing from the patient's perspective. These instruments, the Healing Encounters and Attitudes Lists (HEAL) assess the Patient-Provider Connection, Treatment Expectancy, views of the Healthcare Environment, Positive and Negative Attitudes, Spirituality, and Attitude toward Complementary and Alternative Medicine (CAM). HEAL CAT's, like other PROMIS CATs, are brief, easy to use and understand, and are designed to apply to a broad spectrum of treatments and health conditions. In this project, the investigators aim to 1) evaluate whether HEAL predicts chronic pain treatment outcomes, 2) examine heterogeneity of treatment effects based upon HEAL and PROMIS scores in integrative and conventional medicine settings, and 3) interview patients and their clinicians regarding the utility of HEAL, PROMIS and a Pain Log for enhancing communication. The investigators will administer HEAL CATs and other PROMIS CATs (depression, anxiety, sleep disturbance, fatigue and physical function) to 200 patients who are starting treatment for chronic pain in integrative medicine and conventional medicine settings. Follow-up assessments will be completed 2 and 4 months after baseline testing. The investigators will evaluate factors that may predict which patients judge themselves to be improved, the same, or worsened. Some of the possible factors that may contribute to improvement include HEAL scores, emotional distress, or the preference for CAM or conventional treatment. The investigators are also interested in learning whether patients find the assessments to be clear and useful. A subset of 50 patients and approximately 10 clinicians will complete interviews about the HEAL and PROMIS questions, and about the Pain Log developed by a patient advocacy group partner, the American Chronic Pain Association. By interviewing patients and their healthcare providers, the investigators hope to determine the clarity and acceptability of the HEAL and other assessments, and to learn whether HEAL and PROMIS summaries enhance patient-provider communication in the clinical partnership.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* able to read and understand English
* able to answer questionnaires on a computer
* starting a new treatment for chronic pain or having just started a new treatment within the past month
* expecting to continue their course of treatment

Exclusion Criteria:

* psychotic disorders
* substance abuse by self report

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have ongoing pain (> / = 3 months) who are beginning a treatment for their pain.
Sampling Method: Non-Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2015-02; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol M Greco, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Over a 1 year period, 218 persons beginning treatment for chronic pain at conventional medicine clinics (pain clinics, physical therapy, primary care) (n=105), and integrative medicine centers (n=113) were invited to complete online assessments at 3 time-points: Baseline, 2 month, and 4 month follow-up.
Pre-assignment Details: 9 participants enrolled (completed consent) and did not continue in the study: 2 Integrative / Complementary Alternative Medicine (CAM) and 1 Conventional withdrew after signing consent form; 2 CAM and 4 Conventional did not meet eligibility criteria after signing consent form.
Groups:
- Integrative Medicine Group: Patients receiving chiropractic care, acupuncture, massage therapy, or meditation training for chronic pain
Period: Baseline
Arm/Group | Integrative Medicine Group | Conventional Medicine Group
Started | 109 | 100
Completed | 109 | 100
Not Completed | 0 | 0
Period: 6-8 Weeks
Arm/Group | Integrative Medicine Group | Conventional Medicine Group
Started | 105 (4 CAM participants not eligible to complete follow ups because they did not continue treatment.) | 98 (2 Con. participants not eligible to complete follow ups because they did not continue treatment.)
Completed | 95 | 97
Not Completed | 10 | 1
Not completed — Missed 6-8 week, eligible for 16 week | 10 | 1
Period: 16 Weeks
Arm/Group | Integrative Medicine Group | Conventional Medicine Group
Started | 105 (10 CAM participants Missed 6-8 week but are eligible for 16 week) | 98 (1 Conv. participant Missed 6-8 week but was eligible for 16 week)
Completed | 100 | 96
Not Completed | 5 | 2
Not completed — Completed 6-8 week, missed 16 week | 2 | 2
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Integrative Medicine Group | Conventional Medicine Group | Total
Number analyzed (Participants) | 109 | 100 | 209
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (14.5) | 49.5 (15.0) | 47.5 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 75 | 157
  Male | 27 | 25 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 3 | 14
  Not Hispanic or Latino | 97 | 97 | 194
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 12 | 24 | 36
  White | 87 | 72 | 159
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 2 | 0 | 2
Education [Count of Participants; unit: Participants]
  Less than 4-year degree | 53 | 47 | 100
  Greater than or equal to 4-year degree | 55 | 53 | 108
  Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: PROMIS Pain Intensity
Description: PROMIS Pain Intensity is a three item scale measuring the severity of pain at its worst (past week), average (past week), and current level using a five-point Likert-type scale (i.e., no pain=1, mild=2, moderate=3, severe=4, very severe=5). Scores on the 3 items are summed to create a raw score, which can range from 3 to 15. The raw score is converted to a T-score metric in which 50 is the mean of the relevant reference population and 10 is the standard deviation (SD) of that population.(see http://www.healthmeasures.net/promis-scoring-manuals for details ).
Time Frame: 6-8 weeks
Measure: Mean (Standard Deviation); unit: T-score metric
Arm/Group | Integrative Medicine Group | Conventional Medicine Group
Number analyzed (Participants) | 105 | 98
T-score metric | 50.1 (6.6) | 52.9 (6.2)

2. Primary Outcome: PROMIS Pain Interference
Description: Computerized adaptive test measuring interference of pain in everyday functioning using five-point Likert-type scales with two types or response options (i.e., "not at all"=1, "a little bit"=2, "somewhat"=3, "quite a bit"=4, "very much"=5, and "never"=1, "rarely"=2, "sometimes"=3, "often"=4, "always"=5). Scores on the items are summed to create a raw score. The raw score is converted to a T-score metric in which 50 is the mean of the relevant reference population and 10 is the standard deviation (SD) of that population.(see http://www.healthmeasures.net for details of CAT administration and scoring).
Time Frame: 6-8 weeks
Measure: Mean (Standard Deviation); unit: T-score metric
Arm/Group | Integrative Medicine Group | Conventional Medicine Group
Number analyzed (Participants) | 109 | 100
T-score metric | 59.4 (8.1) | 63.1 (6.6)

3. Secondary Outcome: Clinical Global Impression of Change (CGI)
Description: Patient's rating of current symptom level compared to baseline assessment using a five-point bipolar scale: Much better(2), Somewhat better(1), No change(0), Somewhat worse(-1), Much worse(-2)
Time Frame: 6-8 weeks
Measure: Number; unit: participants
Arm/Group | Integrative Medicine Group | Conventional Medicine Group
Number analyzed (Participants) | 109 | 100
participants
  Much better | 16 | 9
  Better | 46 | 51
  No change | 20 | 23
  Somewhat worse | 4 | 10
  Much worse | 1 | 2
  Missing | 22 | 5

ADVERSE EVENTS:
Time Frame: 6 - 8 weeks
Arm/Group | Integrative Medicine Group | Conventional Medicine Group
All-Cause Mortality (participants affected / at risk) | 0/109 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/109 | 0/100
Other Adverse Events (participants affected / at risk) | 0/109 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes